CLINICAL TRIAL: NCT05873114
Title: Comparison of Effects of Muscle Energy Technique (MET) vs Mobilization in Management of Post-partum Backache in Females With Normal Vaginal Delivery (NVD) and Cesarean Section Delivery
Brief Title: Comparison of MET vs Mobilization in Management of Post-partum Backache in Females (NVD) and Cesarean Section Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/540
Record Dates: First submitted 2023-03-18; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Lipid Mobilization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle Energy Technique (MET) (Experimental)
  Interventions: Diagnostic Test: Muscle Energy Technique (MET)
- Mobilization (Other)
  Interventions: Diagnostic Test: Mobilization

INTERVENTIONS:
Diagnostic Test: Mobilization — Effects of Mobilization in Management of Post-partum Backache in Females With Normal Vaginal Delivery (NVD) and Cesarean Section Delivery
  Arms: Mobilization
Diagnostic Test: Muscle Energy Technique (MET) — Effects of Muscle Energy Technique (MET) in Management of Post-partum Backache in Females With Normal Vaginal Delivery (NVD) and Cesarean Section Delivery
  Arms: Muscle Energy Technique (MET)

SUMMARY:
Effectiveness Comparison of Effects of Muscle Energy Technique (MET) vs Mobilization in Management of Post-partum Backache in Females With Normal Vaginal Delivery (NVD) and Cesarean Section Delivery

ELIGIBILITY:
Inclusion Criteria:

* Subjects with age group 20 to 40 year.
* low back pain and disability after normal vaginal delivery or c-section delivery will be included.

Exclusion Criteria:

* Subjects who had neurological deficit.
* spinal tumors, scoliosis
* underwent spinal surgery
* prolapsed intervertebral disc with or without radiculopathy will be excluded.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
NPSR | 6 Months
  Numeric pain rating scale
Owestry | 6 Months
  Owestry low back pain disability questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudary Muhammad Akram Teaching Hospital, Azra Naheed Medical College, Superior University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No